CLINICAL TRIAL: NCT00860886
Title: Premenopausal Hormone Concentrations in a Population of Women at Very Low Risk of Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909078; 09-C-N078
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Menopause; Normal Physiology
Keywords: Mongolia; Asia; GROWTH FACTORS; Hormones; Premenopausal; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — sera, urine

GROUPS / COHORTS (2):
- 1: Mongolian Women
- 2: Women in other parts of the world other than Mongolia.

SUMMARY:
Background:

* Incidence of breast cancer is very low in Mongolia (6.6/100,000), especially in rural areas. Over the past 15 years, there has been considerable economic growth in Mongolia, resulting in migration to urban centers such as the capital, Ulaanbaatar, from areas with nomadic or semi-nomadic lifestyles. This recent migration offers an opportunity to study the endocrine profiles of premenopausal women as they acculturate to a more Western lifestyle.

Objectives:

* To obtain new data on premenopausal endocrine and growth factor concentrations to assess possible variations by migration status within Ulaanbaatar; that is, to compare women who have been living in Ulaanbaatar for the longest period of time with those who have recently moved to Ulaanbaatar.
* To compare data from Mongolia with data from the United States (and possibly China), where women are at higher risk of breast cancer.

Eligibility:

* A sample of 375 premenopausal women will be drawn from a larger sample of mothers whose children are participating in a study conducted by Harvard Medical School. Only mothers of girls will be included in this cross-sectional study. Women ages 25 44 years who are not pregnant or breastfeeding are eligible.

Design:

* A total of 30 ml (three 10 ml samples) of whole blood will be collected. Women will be asked to provide a spot urine sample. These samples will be sent periodically to the NCI biorespository during the course of the study for testing. A portion of a sample for each participant will be kept in Ulaanbaatar in case of problems in delivery to the United States.
* The following hormones will be evaluated: testosterone, androstenedione, dehydroepiandrosterone (DHEA), DHEA-sulfate, estrone, estradiol, estriol, progesterone, prolactin, placental lactogen, IGF-1 and IGFBP-3, VEGF, soluble endoglin, and possibly other angiogenic proteins.
* Socioeconomic status and medical and lifestyle information will be assessed by questionnaire, including ethnicity, occupation, education, and migration status (e.g., whether she moved from a rural area and time since migration). Breast cancer risk factors such as age at first pregnancy, age at first menstruation, gravidity (total number of pregnancies), parity (total number of childbirths), smoking status, alcohol use, and dietary intake will also be determined. (These questionnaires will have been pilot tested and revised before the start of this study.) The Global Physical Activity Questionnaire, developed by the World Health Organization, will assess physical activity.
* Mean and median premenopausal hormone concentrations of previously collected blood samples from women in the United States who are at high breast cancer risk will be compared with the Mongolian samples. In addition, Chinese data will be compared if available.

DETAILED DESCRIPTION:
There are striking differences in breast cancer incidence rates between Asian and North American and Western European populations, but within Asia variation is also wide. Incidence in Mongolia is one of the lowest in the world (6.6/100,000) while China, its neighbor to the south, has about three times this rate (18.7/100,000). Furthermore, rates appear higher in urban than in rural areas in Mongolia. Over the last decade and a half Mongolia has experienced profound economic changes resulting in mass migration from a nomadic or semi-nomadic existence to a more western lifestyle in the capital city of Ulaanbaatar, and some back migration to rural areas. Together with the contrast in exposures between traditional and urban settings, migration presents the opportunity to study women as they acculturate to a more western lifestyle.

We propose collecting blood and urine samples from premenopausal Mongolian women living in UlaanBaatar, the capital of Mongolia, to describe concentrations of several steroid hormones and growth factors that play a role in breast cancer development. The purpose of the study is to assess whether endocrine profile differs by degree of Western acculturation among those who have recently migrated to the capital. Subjects will be recruited among mothers of girls participating in a study of milk consumption and hormonal status presently being conducted by our colleagues at Harvard Medical School. In addition to the blood draw and urine collection, participants will have their height and weight measured and will complete a questionnaire on reproductive and medical history, migration status and lifestyle factors. Premenopausal blood samples with accompanying information on medical history and lifestyle factors from women participating in Project Viva in Boston, Massachusetts will provide a comparison group of US women at high breast cancer risk.

In general, Asian countries have been treated as one entity and the substantial variation in breast cancer incidence among the countries that make up this large geographic area has not been addressed. This variation among Asian countries may provide further opportunity for hypothesis generating as we seek to determine what factors explain differences in breast cancer rates between populations. Studies of a range of biological parameters in premenopausal women among different racial/ethnic populations with varying breast cancer incidence would be informative.

ELIGIBILITY:
Participants will be drawn from a group of mothers whose children are participating in a study that will be conducted by our colleagues at Harvard Medical School. The Harvard study is a randomized trial among 750 3rd grade children (aged 9-11) to determine the impact of various types of vitamin D fortified and unfortified milk and vitamin D supplements on levels of 25(OHD), growth hormone, and IGF-1. Children in this study will be recruited at eleven primary schools in Ulaanbaatar. The trial will run from January through March 2009 and will include 375 girls; we estimate that their mothers will be roughly 30-45 years of age, and few will be pregnant.

We plan to recruit participants for our study at the time of the baseline blood draw in their daughters. Women ages 25-44 are eligible who are not pregnant or breastfeeding.

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women (ages 25-44)in Mongolia. These women were mothers of children attending several schools in Ulanbaatar (the capital).
Sampling Method: Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2009-03-02 (Actual); Primary Completion 2009-04-15 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
hormone measurements | cross-sectional
  compare hormone measurements of Mongolian women with those of women in other parts of the world.

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Hoover, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Health Sciences University of Mongolia, Ulaanbaatar, Mongolia

REFERENCES:
- [Background] Bernstein L, Yuan JM, Ross RK, Pike MC, Hanisch R, Lobo R, Stanczyk F, Gao YT, Henderson BE. Serum hormone levels in pre-menopausal Chinese women in Shanghai and white women in Los Angeles: results from two breast cancer case-control studies. Cancer Causes Control. 1990 Jul;1(1):51-8. doi: 10.1007/BF00053183. PMID 2102277
- [Background] Bolelli G, Muti P, Micheli A, Sciajno R, Franceschetti F, Krogh V, Pisani P, Berrino F. Validity for epidemiological studies of long-term cryoconservation of steroid and protein hormones in serum and plasma. Cancer Epidemiol Biomarkers Prev. 1995 Jul-Aug;4(5):509-13. PMID 7549807
- [Background] Falk RT, Fears TR, Hoover RN, Pike MC, Wu AH, Nomura AM, Kolonel LN, West DW, Ziegler RG. Does place of birth influence endogenous hormone levels in Asian-American women? Br J Cancer. 2002 Jul 1;87(1):54-60. doi: 10.1038/sj.bjc.6600339. PMID 12085256